CLINICAL TRIAL: NCT01313494
Title: A 6-month, Double-blind, Randomised, Multicenter, Multinational Trial to Investigate the Effect of 500 µg Roflumilast Tablets Once Daily Versus Placebo on Pulmonary Function in Patients With COPD. The ACROSS Trial
Brief Title: A Chronic Obstructive Pulmonary Disease (COPD) Trial Investigating Roflumilast on Safety and Effectiveness in China, Hong Kong and Singapore:
Acronym: ACROSS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RO-2455-301-RD; U1111-1133-6304 (Registry Identifier: WHO)
Record Dates: First submitted 2011-03-03; First posted 2011-03-11 (Estimated); Results first posted 2013-08-02 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2016-09

CONDITIONS: COPD
Keywords: COPD; Roflumilast; FEV1; China
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Roflumilast; Albuterol

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Roflumilast (Experimental): Roflumilast 500 μg, tablet, oral, once daily for up to 24 weeks.
  Interventions: Drug: Roflumilast; Drug: Salbutamol
- Placebo (Placebo Comparator): Placebo to roflumilast, tablet, oral, once daily for up to 24 weeks.
  Interventions: Drug: Placebo; Drug: Salbutamol

INTERVENTIONS:
Drug: Roflumilast — Roflumilast tablets
  Arms: Roflumilast
Drug: Placebo — Placebo tablets
  Arms: Placebo
Drug: Salbutamol — Salbutamol (given by MDI and spacer) used as rescue medication on an ass needed basis throughout the trial, and was used for post-bronchodilator spirometry tests at all study visits.

SUMMARY:
The aim of this trial is to determine the efficacy, safety and tolerability of 500 µg Roflumilast tablets once daily in patients with COPD in China, Hong Kong, and Singapore.

ELIGIBILITY:
Main Inclusion Criteria:

* Willingness to sign a written informed consent
* Chronic obstructive pulmonary disease (COPD) according to Global Initiative for Chronic Obstructive Lung Disease (GOLD) guidelines 2009
* Chinese or Malay or Indian ethnicity
* History of chronic obstructive pulmonary disease symptoms for at least 12 months prior to baseline visit V0
* Forced expiratory volume in the first second/ Forced vital capacity (FEV1/FVC) ratio (post-bronchodilator) < 70%
* Forced expiratory volume in the first second (FEV1) (post-bronchodilator) < 50 % of predicted
* Former smoker (defined as: smoking cessation at least one year ago) or current smoker both with a smoking history of at least 10 pack years

Main Exclusion Criteria:

* Moderate or severe COPD exacerbation and/or COPD exacerbations treated with antibiotics not stopped at V0
* Lower respiratory tract infection not resolved 4 weeks prior to the baseline visit V0
* History of asthma diagnosis in patients < 40 years of age or relevant lung disease other than COPD
* Current participation in a pulmonary rehabilitation program or completion of a pulmonary rehabilitation program within 3 months preceding the baseline visit V0
* Known alpha-1-antitrypsin deficiency

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 626 (Actual)
Dates: Start 2011-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (15):
- China (13):
  - Beijing
  - Changsha
  - Chengdu
  - Chongqing
  - Fuzhou
  - Guangzhou
  - Hangzhou
  - Nanjing
  - Nanning
  - Qingdao
  - Shanghai
  - Shenyang
  - Shijiazhuang
- Hong Kong, Hong Kong
- Singapore, Singapore

REFERENCES:
- [Derived] Zheng J, Yang J, Zhou X, Zhao L, Hui F, Wang H, Bai C, Chen P, Li H, Kang J, Brose M, Richard F, Goehring UM, Zhong N. Roflumilast for the treatment of COPD in an Asian population: a randomized, double-blind, parallel-group study. Chest. 2014 Jan;145(1):44-52. doi: 10.1378/chest.13-1252. PMID 24135893

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 43 investigative sites in mainland China, Hong Kong and Singapore from 04 Mar 2011 to 16 May 2012.
Pre-assignment Details: Participants with a diagnosis of chronic obstructive pulmonary disease (COPD) were randomized in 1 of 2 treatment groups (placebo and roflumilast 500 μg once daily).
Period: Overall Study
Arm/Group | Roflumilast | Placebo
Started | 313 | 313
Safety Set | 315 (2 patients in the placebo arm were misallocated and may have received roflumilast in error.) | 311 (2 patients in the placebo arm were misallocated and may have received roflumilast in error.)
Completed | 246 | 263
Not Completed | 67 | 50

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Roflumilast | Placebo | Total
Number analyzed (Participants) | 313 | 313 | 626
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.2 (8.76) | 64.0 (8.27) | 64.1 (8.51)
Gender [Count of Participants; unit: Participants]
  Female | 30 | 27 | 57
  Male | 283 | 286 | 569
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 313 | 313 | 626
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: cm] | 166.2 (7.27) | 165.9 (7.12) | 166.1 (7.20)
Weight [Mean (Standard Deviation); unit: kg] | 60.4 (11.00) | 61.8 (10.54) | 61.1 (10.78)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 21.8 (3.42) | 22.4 (3.43) | 22.1 (3.44)
Chronic obstructive pulmonary disease (COPD) severity [Number; unit: Participants] — COPD severity was classified according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD) Guideline (2009) as: - Very severe COPD: baseline post-bronchodilator FEV1 %predicted < 30% - Severe COPD: baseline post-bronchodilator FEV1 %predicted ≥ 30% to < 50% - Moderate COPD: baseline post-bronchodilator FEV1 %predicted ≥ 50% to < 80% - Mild COPD: baseline post-bronchodilator FEV1 %predicted ≥ 80%.
  Participants
    Mild | 1 | 1 | 2
    Moderate | 28 | 16 | 44
    Severe | 196 | 204 | 400
    Very severe | 88 | 92 | 180
COPD disease characteristics [Number; unit: Participants]
  Predominantly chronic bronchitis | 56 | 61 | 117
  Combined emphysema and chronic bronchitis | 217 | 216 | 433
  Predominantly emphysema | 40 | 36 | 76
Smoking status [Number; unit: Participants]
  Former smoker | 238 | 221 | 459
  Current smoker | 75 | 92 | 167
Cigarette pack years [Mean (Standard Deviation); unit: pack years] | 37.2 (21.18) | 37.5 (23.00) | 37.4 (22.09)
Pre-bronchodilator forced expiratory volume in the first second (FEV1) [Mean (Standard Deviation); unit: Liters] | 0.8 (0.31) | 0.8 (0.24) | 0.8 (0.28)
Post-bronchodilator FEV1 [Mean (Standard Deviation); unit: Liters] | 1.0 (0.35) | 0.9 (0.27) | 0.9 (0.31)
Pre-bronchodilator FEV1 predicted [Mean (Standard Deviation); unit: Percent of predicted] | 32.7 (10.23) | 32.7 (9.00) | 32.7 (9.63)
Post-bronchodilator FEV1 predicted [Mean (Standard Deviation); unit: Percent of predicted] | 36.8 (11.42) | 36.4 (10.13) | 36.6 (10.79)
FEV1 reversibility increase [Mean (Standard Deviation); unit: mL] | 108.4 (110.83) | 94.8 (104.71) | 101.6 (107.94)
FEV1 reversibility % increase [Mean (Standard Deviation); unit: Percent reversibility] — FEV reversibility (%) = (post-bronchodilator FEV minus pre-bronchodilator FEV) / pre-bronchodilator FEV * 100.
  Percent reversibility | 13.6 (15.29) | 11.8 (13.15) | 12.7 (14.27)
Post-bronchodilator FEV1/forced vital capacity (FVC) [Mean (Standard Deviation); unit: FEV1/FVC percent] — Calculated as FEV1/FVC * 100
  FEV1/FVC percent | 35.8 (9.69) | 35.3 (8.92) | 35.5 (9.31)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Pre-bronchodilator Forced Expiratory Volume in First Second (FEV1)
Description: FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation. Pulmonary function testing was performed using centralized spirometry prior to taking study medication. Change from baseline over 24 weeks of treatment was calculated from a repeated measures analysis of covariance (ANCOVA) model with treatment, baseline value of pre-bronchodilator FEV1, time and a treatment-by-time interaction as independent variables.
Time Frame: Baseline to Week 24
Population: Intent-to-treat population included all randomly assigned patients who took at least 1 dose of trial treatment after randomization. Patients were assigned to the treatment group based on the treatment to which they were randomly assigned. Only patients with available data at Baseline and with at least 1 post-baseline measurement are included.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 295 | 305
liters | 0.049 (0.009) | -0.022 (0.009)
Statistical Analysis 1: Comparison: Roflumilast vs Placebo; The primary endpoint was tested in a confirmatory manner with a 2-sided significance level of 5%; Test type: Superiority or Other; p < 0.0001, Repeated measures ANCOVA; Independent variables: treatment, baseline value of pre-bronchodilator FEV1, time and a treatment-by-time interaction; LSM Difference = 0.071, 95% CI 2-sided [0.046 to 0.095], Standard Error of Mean 0.012

2. Secondary Outcome: Change From Baseline in Post-bronchodilator FEV1
Description: FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation. Pulmonary function testing was performed using centralized spirometry prior to taking study medication. Post-bronchodilator measurements were taken 30 minutes after four inhalations of 100 μg salbutamol. Change from baseline over 24 weeks of treatment was calculated from a repeated measures analysis of covariance (ANCOVA) model with treatment, baseline value of post-bronchodilator FEV1, time and a treatment-by-time interaction as independent variables.
Time Frame: Baseline to Week 24
Population: Intent-to-treat population with available data.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 295 | 305
liters | 0.045 (0.009) | -0.023 (0.009)

3. Secondary Outcome: Change From Baseline in Pre-bronchodilator Forced Vital Capacity (FVC)
Description: Vital capacity is the amount of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. Pulmonary function testing was performed using centralized spirometry prior to taking study medication. Change from baseline over 24 weeks of treatment was calculated from a repeated measures analysis of covariance (ANCOVA) model with treatment, baseline value, time and a treatment-by-time interaction as independent variables.
Time Frame: Baseline to Week 24
Population: Intent-to-treat population with available data.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 295 | 305
liters | 0.100 (0.017) | -0.009 (0.017)

4. Secondary Outcome: Change From Baseline in Post-bronchodilator Forced Vital Capacity (FVC)
Description: Vital capacity is the amount of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. Pulmonary function testing was performed using centralized spirometry prior to taking study medication. Post-bronchodilator measurements were taken 30 minutes after four inhalations of 100 μg salbutamol. Change from baseline over 24 weeks of treatment was calculated from a repeated measures analysis of covariance (ANCOVA) model with treatment, baseline value, time and a treatment-by-time interaction as independent variables.
Time Frame: Baseline to Week 24
Population: Intent-to-treat population with available data.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 295 | 305
liters | 0.094 (0.017) | -0.007 (0.016)

5. Secondary Outcome: Change From Baseline in Pre-bronchodilator Forced Expiratory Flow 25-75%
Description: Forced expiratory flow 25-75% (FEF25-75%) is the flow (or speed) of air coming out of the lung during the middle half of a forced expiration. Pulmonary function testing was performed using centralized spirometry prior to taking study medication. Change from baseline over 24 weeks of treatment was calculated from a repeated measures analysis of covariance (ANCOVA) model with treatment, baseline value, time and a treatment-by-time interaction as independent variables.
Time Frame: Baseline to Week 24
Population: Intent-to-treat population with available data.
Measure: Least Squares Mean (Standard Error); unit: liters/second
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 295 | 305
liters/second | 0.023 (0.005) | -0.010 (0.005)

6. Secondary Outcome: Change From Baseline in Post-bronchodilator Forced Expiratory Flow 25-75%
Description: Forced expiratory flow 25-75% (FEF25-75%) is the flow (or speed) of air coming out of the lung during the middle half of a forced expiration. Pulmonary function testing was performed using centralized spirometry prior to taking study medication. Post-bronchodilator measurements were taken 30 minutes after four inhalations of 100 μg salbutamol. Change from baseline over 24 weeks of treatment was calculated from a repeated measures analysis of covariance (ANCOVA) model with treatment, baseline value, time and a treatment-by-time interaction as independent variables.
Time Frame: Baseline to Week 24
Population: Intent-to-treat population with available data.
Measure: Least Squares Mean (Standard Error); unit: liters/second
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 295 | 305
liters/second | 0.022 (0.005) | -0.008 (0.005)

7. Secondary Outcome: Change From Baseline in Pre-bronchodilator Forced Expiratory Volume in First Three Seconds (FEV3)
Description: FEV3 is the amount of air which can be forcibly exhaled from the lungs in the first three seconds of a forced exhalation. Pulmonary function testing was performed using centralized spirometry prior to taking study medication. Change from baseline over 24 weeks of treatment was calculated from a repeated measures analysis of covariance (ANCOVA) model with treatment, baseline value of pre-bronchodilator FEV3, time and a treatment-by-time interaction as independent variables.
Time Frame: Baseline to Week 24
Population: Intent-to-treat population with available data.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 295 | 305
liters | 0.072 (0.012) | -0.030 (0.012)

8. Secondary Outcome: Change From Baseline in Post-bronchodilator Forced Expiratory Volume in First Three Seconds (FEV3)
Description: FEV3 is the amount of air which can be forcibly exhaled from the lungs in the first three seconds of a forced exhalation. Pulmonary function testing was performed using centralized spirometry prior to taking study medication. Post-bronchodilator measurements were taken 30 minutes after four inhalations of 100 μg salbutamol. Change from baseline over 24 weeks of treatment was calculated from a repeated measures analysis of covariance (ANCOVA) model with treatment, baseline value of post-bronchodilator FEV3, time and a treatment-by-time interaction as independent variables.
Time Frame: Baseline to Week 24
Population: Intent-to-treat population with available data.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 295 | 305
liters | 0.064 (0.012) | -0.030 (0.011)

9. Secondary Outcome: Change From Baseline in Pre-bronchodilator Forced Expiratory Volume in First Six Seconds (FEV6)
Description: FEV6 is the amount of air which can be forcibly exhaled from the lungs in the first six seconds of a forced exhalation. Pulmonary function testing was performed using centralized spirometry prior to taking study medication. Change from baseline over 24 weeks of treatment was calculated from a repeated measures analysis of covariance (ANCOVA) model with treatment, baseline value of pre-bronchodilator FEV6, time and a treatment-by-time interaction as independent variables.
Time Frame: Baseline to Week 24
Population: Intent-to-treat population with available data.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 295 | 305
liters | 0.084 (0.014) | -0.031 (0.014)

10. Secondary Outcome: Change From Baseline in Post-bronchodilator Forced Expiratory Volume in First Six Seconds (FEV6)
Description: FEV6 is the amount of air which can be forcibly exhaled from the lungs in the first three seconds of a forced exhalation. Pulmonary function testing was performed using centralized spirometry prior to taking study medication. Post-bronchodilator measurements were taken 30 minutes after four inhalations of 100 μg salbutamol. Change from baseline over 24 weeks of treatment was calculated from a repeated measures analysis of covariance (ANCOVA) model with treatment, baseline value of post-bronchodilator FEV6, time and a treatment-by-time interaction as independent variables.
Time Frame: Baseline to Week 24
Population: Intent-to-treat population with available data.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 295 | 304
liters | 0.078 (0.013) | -0.032 (0.013)

11. Secondary Outcome: Change From Baseline in Pre-bronchodilator Peak Expiratory Flow Rate (PEF)
Description: PEF is the maximal flow (or speed) achieved during the maximally forced expiration initiated at full inspiration. Pulmonary function testing was performed using centralized spirometry prior to taking study medication. Change from baseline over 24 weeks of treatment was calculated from a repeated measures analysis of covariance (ANCOVA) model with treatment, baseline value, time and a treatment-by-time interaction as independent variables.
Time Frame: Baseline to Week 24
Population: Intent-to-treat population with available data.
Measure: Least Squares Mean (Standard Error); unit: liters/minute
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 295 | 305
liters/minute | 0.096 (0.027) | -0.036 (0.026)

12. Secondary Outcome: Change From Baseline in Post-bronchodilator Peak Expiratory Flow Rate (PEF)
Description: PEF is the maximal flow (or speed) achieved during the maximally forced expiration initiated at full inspiration. Pulmonary function testing was performed using centralized spirometry prior to taking study medication. Post-bronchodilator measurements were taken 30 minutes after four inhalations of 100 μg salbutamol. Change from baseline over 24 weeks of treatment was calculated from a repeated measures analysis of covariance (ANCOVA) model with treatment, baseline value, time and a treatment-by-time interaction as independent variables.
Time Frame: Baseline to Week 24
Population: Intent-to-treat population with available data.
Measure: Least Squares Mean (Standard Error); unit: liters/minute
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 295 | 305
liters/minute | 0.099 (0.027) | -0.030 (0.027)

13. Secondary Outcome: Change From Baseline in Pre-bronchodilator Ratio of Forced Expiratory Volume After 1 Second to Forced Vital Capacity
Description: The FEV1/FVC ratio represents the percentage of vital capacity expelled from the lungs during the first second of a forced exhalation. Pulmonary function testing was performed using centralized spirometry prior to taking study medication.
Time Frame: Baseline and Week 24
Population: Intent-to-treat population with available data; last observation carried forward (LOCF) was used.
Measure: Median (Full Range); unit: percent FEV1/FVC
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 295 | 305
percent FEV1/FVC | -0.570 (4.5667) [-14.32 to 28.35] | -1.370 (4.9968) [-19.81 to 27.36]

14. Secondary Outcome: Change From Baseline in Post-bronchodilator Ratio of Forced Expiratory Volume After 1 Second to Forced Vital Capacity
Description: The FEV1/FVC ratio represents the percentage of vital capacity expelled from the lungs during the first second of a forced exhalation. Pulmonary function testing was performed using centralized spirometry prior to taking study medication. Post-bronchodilator measurements were taken 30 minutes after four inhalations of 100 μg salbutamol.
Time Frame: Baseline and Week 24
Population: Intent-to-treat population with available data; last observation carried forward (LOCF) was used.
Measure: Median (Full Range); unit: percent FEV1/FVC
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 295 | 305
percent FEV1/FVC | -0.320 (4.5400) [-16.38 to 18.30] | -0.940 (5.1677) [-23.53 to 33.77]

15. Secondary Outcome: Change From Baseline in Pre-bronchodilator Ratio of Forced Expiratory Volume After 1 Second to Forced Expiratory Volume After 6 Seconds
Description: The FEV1/FEV6 ratio represents the percentage of the volume of air expired in the first six seconds that is expelled from the lungs during the first second of a forced exhalation. Pulmonary function testing was performed using centralized spirometry prior to taking study medication.
Time Frame: Baseline and Week 24
Population: Intent-to-treat population with available data; last observation carried forward (LOCF) was used.
Measure: Median (Full Range); unit: percentage of FEV1/FEV6
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 295 | 305
percentage of FEV1/FEV6 | -0.210 (3.9213) [-14.05 to 27.48] | -0.950 (3.9173) [-17.09 to 21.03]

16. Secondary Outcome: Change From Baseline in Post-bronchodilator Ratio of Forced Expiratory Volume After 1 Second to Forced Expiratory Volume After 6 Seconds
Description: The FEV1/FEV6 ratio represents the percentage of the volume of air expired in the first six seconds that is expelled from the lungs during the first second of a forced exhalation. Pulmonary function testing was performed using centralized spirometry prior to taking study medication. Post-bronchodilator measurements were taken 30 minutes after four inhalations of 100 μg salbutamol.
Time Frame: Baseline and Week 24
Population: Intent-to-treat population with available data; last observation carried forward (LOCF) was used.
Measure: Mean (Full Range); unit: percentage of FEV1/FEV6
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 295 | 304
percentage of FEV1/FEV6 | -0.340 (3.7240) [-25.56 to 17.08] | -0.420 (4.1957) [-20.53 to 25.55]

17. Secondary Outcome: Change From Baseline in COPD Symptom Scores
Description: Symptoms of chronic bronchitis with respect to cough and sputum production were assessed daily by the patient and recorded in a diary. Symptoms were assessed on a 4-point scale as follows: Cough: 0: no cough; 1: mild cough (at some time during the day); 2: moderate cough (regularly during the day); 3: severe cough (never free of cough or feeling free of need to cough). Sputum production: 0: no sputum production (unnoticeable); 1: mild sputum production (noticeable as a problem); 2: moderate sputum production (frequent inconvenience); 3: severe sputum production (constant problem). Change from Baseline is reported for cough and sputum separately, and for the sum of the 2 scores (range 0 - 6). Least squares means (LSM) are from a repeated measures ANCOVA model with treatment, baseline value, time and a treatment-by-time interaction as independent variables.
Time Frame: Baseline to Week 24
Population: Intent-to-treat population with available data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 284 | 299
units on a scale
  Score Sum (n=282, 296) | 0.013 (0.054) | 0.064 (0.053)
  Cough (n=284, 299) | -0.019 (0.029) | 0.036 (0.028)
  Sputum (n=284, 296) | 0.035 (0.030) | 0.037 (0.029)

18. Secondary Outcome: Change From Baseline in Use of Rescue Medication
Description: Salbutamol (given by metered dose inhaler and spacer) was used as rescue medication according to the individual needs of a patient. Each use was documented in the patient's paper diary. Least squares means (LSM) are from a repeated measures ANCOVA model with treatment, baseline value, time and a treatment-by-time interaction as independent variables.
Time Frame: Baseline to Week 24
Population: Intent-to-treat population with available data.
Measure: Least Squares Mean (Standard Error); unit: puffs/day
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 286 | 293
puffs/day | -0.485 (0.134) | -0.518 (0.131)

19. Secondary Outcome: Transition Dyspnoea Index (TDI) Total Score at Week 24
Description: The TDI is a recognized questionnaire to measure dyspnoea (shortness of breath) in patients with COPD. Questions from the TDI were used to assess the 3 components: "change in functional impairment", "change in magnitude of task" and "change in magnitude of effort". Transitions or changes from baseline are rated from -3 (major deterioration) to +3 (major improvement), and summed to give a total score ranging from -9 to +9. Least squares means (LSM) are from a repeated measures ANCOVA model with treatment, baseline value, time and a treatment-by-time interaction as independent variables.
Time Frame: Baseline to Week 24
Population: Intent-to-treat population with available data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 299 | 305
units on a scale | 1.335 (0.124) | 1.396 (0.122)

20. Secondary Outcome: Percentage of Participants With Moderate or Severe COPD Exacerbations
Description: A COPD exacerbation is an event characterised by a worsening in the patient's baseline dyspnoea, or cough and/or sputum beyond day-to-day variability sufficient to warrant a change in management, and may be accompanied by increased wheeze, chest tightness, purulent sputum and symptoms of cold and/or fatigue. COPD exacerbations were categorized as follows: - Severe: Requiring hospitalization and/or leading to death; - Moderate: Requiring oral or parenteral glucocorticosteroid therapy.
Time Frame: 24 weeks
Population: Intent-to-treat
Measure: Number; unit: percentage of participants
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 313 | 313
percentage of participants
  No exacerbations | 81.8 | 84.7
  One exacerbation | 15.0 | 12.8
  Two exacerbations | 2.6 | 1.9
  Three exacerbations | 0.6 | 0.6

21. Secondary Outcome: Mean Rate of Moderate or Severe COPD Exacerbations Per Patient Per Year
Description: The mean rate of COPD exacerbations per patient per year rate = (number of exacerbations per treatment group/time to study withdrawal per treatment group) * 365. COPD exacerbations were categorized as follows: - Severe: Requiring hospitalization and/or leading to death; - Moderate: Requiring oral or parenteral glucocorticosteroid therapy.
Time Frame: 24 weeks
Population: Intent-to-treat
Measure: Number; unit: exacerbations per patient per year
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 313 | 313
exacerbations per patient per year | 0.55 | 0.44

22. Secondary Outcome: Time to Onset of First Moderate or Severe COPD Exacerbation
Description: Time to onset of a COPD exacerbation is defined as onset date of COPD exacerbation - date of first intake of study drug + 1 day. COPD exacerbations were categorized as follows: - Severe: Requiring hospitalization and/or leading to death; - Moderate: Requiring oral or parenteral glucocorticosteroid therapy.
Time Frame: 24 weeks
Population: Intent-to-treat population with at least one moderate or severe exacerbation
Measure: Median (Full Range); unit: days
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 57 | 48
days | 67.0 [3 to 165] | 86.0 [2 to 168]

23. Secondary Outcome: Time to Onset of Second Moderate or Severe COPD Exacerbation
Description: Time to onset of a COPD exacerbation is defined as onset date of COPD exacerbation - date of first intake of study drug + 1 day. At least 10 days between the stop date of an exacerbation and the start date of the following exacerbation was required for these to be be considered as two separate COPD exacerbations. COPD exacerbations were categorized as follows: - Severe: Requiring hospitalization and/or leading to death; - Moderate: Requiring oral or parenteral glucocorticosteroid therapy.
Time Frame: 24 weeks
Population: Intent-to-treat population who experienced a second moderate to severe COPD exacerbation.
Measure: Median (Full Range); unit: days
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 10 | 8
days | 119.5 [50 to 166] | 117.0 [71 to 163]

24. Secondary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence in a clinical trial participant regardless of causal relationship to study drug and regardless whether study drug has been administered. A serious adverse event (SAE) is any untoward medical occurrence or effect that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability / incapacity, is a congenital anomaly / birth defect or is medically important due to other reasons than the above mentioned criteria. A non-serious AE is any AE that does not meet the criteria above. Each AE was assessed by the Investigator as either 'related' or 'not related' to study drug.
Time Frame: 24 weeks
Population: Safety population, all randomized patients who took at least 1 dose of the trial treatment after randomization.
Measure: Number; unit: participants
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 315 | 311
participants
  All AEs | 213 | 196
  Non-serious AEs | 189 | 172
  Serious AEs (including death) | 62 | 48
  Death | 2 | 2
  Serious AEs not including death | 60 | 46
  AEs with suggested relationship to trial treatment | 65 | 18
  AEs leading to withdrawal from the trial | 15 | 2
  AEs not recovered at trial termination | 54 | 45
  AEs with changes in concomitant medication | 164 | 155

ADVERSE EVENTS:
Time Frame: 24 weeks.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Roflumilast | Placebo
Serious Adverse Events (participants affected / at risk) | 62/315 | 48/311
Other Adverse Events (participants affected / at risk) | 143/315 | 133/311
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Roflumilast (N=315) | Placebo (N=311)
Acute myocardial infarction (Cardiac disorders) | 2 | 0
Angina unstable (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 1 | 1
Cor pulmonale chronic (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 1
Colonic polyp (Gastrointestinal disorders) | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Hepatitis B (Hepatobiliary disorders) | 1 | 0
Liver injury (Hepatobiliary disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 1
Herpes zoster infection neurological (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Ureteric dilatation (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 | 1
Epididymitis (Reproductive system and breast disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 44 | 39
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Varicose vein (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Roflumilast (N=315) | Placebo (N=311)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 90 | 89
Nasopharyngitis (Infections and infestations) | 28 | 45
Upper respiratory tract infection (Infections and infestations) | 17 | 18
Diarrhoea (Gastrointestinal disorders) | 21 | 3
Decreased appetite (Metabolism and nutrition disorders) | 19 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.